CLINICAL TRIAL: NCT04282317
Title: Magnetic Resonance Imaging of the Brain and the Upper Gastrointestinal Tract in Healthy Volunteers and Patients With Gastroparesis
Brief Title: Magnetic Resonance Imaging of the Brain and Stomach in Healthy Volunteers and Gastroparesis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Purdue University (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, John M. Wo, Director of GI Motility and Neurogastroenterology Unit, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MRI study; OT2OD023847 (NIH)
Record Dates: First submitted 2019-12-19; First posted 2020-02-24 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Gastroparesis
Keywords: Gastroparesis; functional MRI; Gastric MRI; Brain MRI
MeSH Terms: conditions — Gastroparesis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteer (Other): This arm will enroll healthy volunteers as controls
  Interventions: Other: MRI scan
- Gastroparesis Subjects (Other): This arm will enroll a) patients with gastroparesis from type 1 diabetes and b) patients with gastroparesis from vagus nerve trauma
  Interventions: Other: MRI scan

INTERVENTIONS:
Other: MRI scan — MRI scan

SUMMARY:
The study is to lay the groundwork for non invasive imaging of the GI tract and the brain gut interaction

DETAILED DESCRIPTION:
Magnetic resonance imaging (MRI) produces non-invasive exquisite spatial resolution of internal organs. However, its application to the GI tract has been limited by several challenges. The GI tract has a complex and convoluted geometry. The GI geometry changes slowly over the course of meal digestion, as well as rapidly due to contraction of various compartments of the GI tract. As a person takes natural breaths during MRI, the respiratory motion further complicates the acquisition and analysis of GI images. In addition, different types of meal or nutrients have variable property as image contrast in upper GI MRI. It is difficult to standardize the MRI analysis for accurate and quantitative assessment of gastric emptying, motility, absorption, and secretion, to name a few. In a recently published study by our research collaborators at Purdue University, they have addressed many of these challenges in rodents and are ready to refine and translate their technical solutions to human upper GI MRI.

Functional MRI of the brain has been used to study afferent response in various GI disorders, such as dysphagia, functional dyspepsia, and irritable bowel syndrome.1-3 Brain activity is altered in the emotional response areas, and activity is reduced in the areas associated with top-down modulation of visceral afferent signals.4 However, direct correlation between regional brain activation by functional-MRI and GI motility by meal-contrast MRI is lacking.

The outcome of the proposed research is expected to lay the groundwork for non-invasive imaging of GI anatomy and function and the brain-gut interaction towards better understanding, diagnosis, prevention, and treatment of GI disorders.

ELIGIBILITY:
HEALTHY VOLUNTEERS

Inclusion Criteria:

• Healthy volunteers from 18 to 65 years of age

Exclusion Criteria:

* Contraindication to MR scanning: pregnancy, implanted gastric stimulator, neural stimulator, implanted cardiac pacemaker, auto-defibrillator, cochlear implant, ocular foreign body (e.g. metal shavings), pain pump, insulin pump or any pre-existing eye conditions.
* Presence of gastroparesis symptoms, such as nausea, emesis, early satiety, effortless regurgitation, post-prandial fullness and pain, and/or postprandial epigastric pain.
* Prior diagnosis of the upper GI disorders, including gastroparesis, gastric or duodenal ulcer, gastric outlet obstruction, acute or chronic pancreatitis, large hiatal or paraesophageal hernia, small intestinal bacterial overgrowth, celiac disease, Crohn's disease.
* Prior systemic disorders associated with GI neuromuscular disorder listed in Appendix B.
* Taking medications that can effect GI motility, including opiate, metoclopramide, dopamine agonist for Parkinson or restless leg syndrome, anticholinergics.
* Prior brain or abdominal surgery (except cholecystectomy or appendectomy).
* Prior diagnosis of central nervous system illness, neurological lesion, a psychiatric history, or recurrent migraines that require medication.
* Uncontrolled medical problems, such as hypertension, pulmonary or airway disease, heart failure, or coronary artery disease.
* Allergy to pineapple.
* Presence of dysphagia.
* Unable to give own informed consent.

GASTROPARESIS PATIENTS

Inclusion Criteria:

* Patients with gastroparesis from 18 to 65 years of age.
* Symptoms of gastroparesis of at least 12 weeks duration with varying degrees of nausea, emesis, early satiety, effortless regurgitation, post-prandial fullness and pain, and/or postprandial epigastric pain.
* Abnormal 4-hour gastric emptying scintigraphy within the last 6 months >60% retention at 2 hrs and/or >10% retention at 4 hrs.

Exclusion Criteria:

* Contraindication to MR scanning: pregnancy, implanted gastric stimulator, neural stimulator, implanted cardiac pacemaker, auto-defibrillator, cochlear implant, ocular foreign body (e.g. metal shavings), pain pump, insulin pump or any pre-existing eye conditions.
* Prior diagnosis of the upper GI disorders other than gastroparesis, including gastric or duodenal ulcer, gastric outlet obstruction, acute or chronic pancreatitis, large hiatal or paraesophageal hernia, small intestinal bacterial overgrowth, celiac disease, Crohn's disease .
* Prior brain or abdominal surgery (except cholecystectomy or appendectomy).
* Prior diagnosis of central nervous system illness, neurological lesion, a psychiatric history, or recurrent migraines that require medication.
* Uncontrolled medical problems, such as hypertension, pulmonary or airway disease, heart failure, or coronary artery disease.
* Allergy to pineapple.
* Prior history of dysphagia.
* Unable to give own informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastric peristalsis | Baseline
  Compare 3D gastric peristalsis progression before & after test meals in healthy volunteers and patients with gastroparesis

SECONDARY OUTCOMES:
Contraction frequency | Baseline
  Compare colored 3-D heat map of stomach contraction frequency before & after test meals in healthy volunteers and patients with gastroparesis
Pylorus transit | Baseline
  Compare pylorus mean opening diameter before & after test meals in healthy volunteers and patients with gastroparesis

CONTACTS AND LOCATIONS:
Overall Officials: John M Wo, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States